CLINICAL TRIAL: NCT03979846
Title: A Pilot Assessment of a Digital System for Cancer Patient Symptom Reporting
Brief Title: A Computer-Based System for Symptom Reporting in Patients With Cancer Undergoing Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: 19F.163; JT 13449 (Other: JeffTrial Number); R43MD011210 (NIH)
Record Dates: First submitted 2019-05-28; First posted 2019-06-07 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Caregiver; Malignant Neoplasm
MeSH Terms: conditions — Neoplasms | interventions — Practice Guidelines as Topic; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (usual care, computer-based symptom reporting) (Experimental): Participants receive usual care for 3 weeks, then use a computer based symptom reporting system for 3 weeks. Caregivers may assist patients in the use of the computer based symptoms reporting system.
  Interventions: Other: Best Practice; Other: Computer Application; Other: Questionnaire Administration; Other: Quality-of-Life Assessment
- Arm II (computer-based symptom reporting, usual care) (Experimental): Participants use a computer based symptom reporting system for 3 weeks, then receive usual care for 3 weeks. Caregivers may assist patients in the use of the computer based symptoms reporting system.
  Interventions: Other: Best Practice; Other: Computer Application; Other: Questionnaire Administration; Other: Quality-of-Life Assessment

INTERVENTIONS:
Other: Best Practice — Receive usual care
  Other Names: standard of care; standard therapy
Other: Computer Application — Use computer-based symptom reporting system
  Other Names: Application; application software; computer applicaion
Other: Questionnaire Administration — Ancillary studies
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment

SUMMARY:
This pilot trial studies the usability and usefulness of a computer-based system for reporting symptoms in patients with cancer undergoing treatment. Cancer patients undergoing cancer treatment are not always comfortable contacting the doctor when experiencing symptoms. A computer based platform, where patients can input symptoms, may seem less intrusive than a phone call and may improve patient access to care.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the usability and usefulness of a computer-based system for cancer patient symptom reporting.

SECONDARY OBJECTIVES:

I. To collect preliminary effectiveness data: quality of life outcomes with the Function Assessment of Cancer Therapy - General (FACT-G) and self-efficacy as measured by Chronic Disease Self-Efficacy Scale, Revised (CDSES-R).

OUTLINE: Participants are randomized to 1 of 2 arms.

ARM I: Participants receive usual care for 3 weeks, then use a computer-based symptom reporting system for 3 weeks. Caregivers may assist patients in the use of the computer based symptoms reporting system.

ARM II: Participants use a computer-based symptom reporting system for 3 weeks, then receive usual care for 3 weeks. Caregivers may assist patients in the use of the computer based symptoms reporting system.

After completing study intervention, participants are followed up for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* PATIENT: Active outpatient cancer treatment (chemotherapy, immunotherapy, radiation, and hormonal therapy)
* PATIENT: No clinical evidence of cognitive or psychological impairment.
* PATIENT: Home internet access on computer or phone.
* CAREGIVER: Selected family member or close friend of the cancer patient matching the patient inclusion criteria outlined above.

Exclusion Criteria:

* Inability to provide informed consent.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-03-11 (Actual); Primary Completion 2019-05-29 (Actual); Study Completion 2019-05-29 (Actual)

PRIMARY OUTCOMES:
Usability of the computer-based symptom reporting system | 6 weeks
  Assessed with the System Usability Scale (SUS). The SUS is a 10-item 5-point Likert scale usability measure, scored from 0 (least usable) to 100 (most usable). The mean SUS scores (only during the active cancer treatment) will be computed with the corresponding 90% confidence intervals.
Patient-deemed usefulness of computer-based symptom reporting system | 6 weeks
  Assessed with the Perceived System Usefulness (PSU) scale. The mean PSU scores (only during the active cancer treatment) will be computed with the corresponding 90% confidence intervals.
Effectiveness of the computer-based symptom reporting system (FACT-G) | 6 weeks
  Evaluated using the quality of life outcome Functional Assessment of Cancer Therapy - General (FACT-G) scale. For the FACT-G, the 4 repeated measures (excluding the baseline) will be analyzed in linear mixed effects models with the random effect of user group (patient and caregiver) and fixed effect of period, sequence. The model will be used to compute the 90% confidence intervals for the mean FACT-G on usual care and on the digital system.
Effectiveness of the computer-based symptom reporting system (CDSES-R) | 6 weeks
  Evaluated using the self-efficacy Chronic Disease Self-Efficacy Scale, Revised (CDSES-R) scale. For the CDSES-R, the 4 repeated measures (excluding the baseline) will be analyzed in linear mixed effects models with the random effect of user group (patient and caregiver) and fixed effect of period, sequence. The model will be used to compute the 90% confidence intervals for the mean CDSES-R on usual care and on the digital system.

CONTACTS AND LOCATIONS:
Overall Officials: Ana Maria Lopez, MD, Principal Investigator — Sidney Kimmel Cancer Center at Thomas Jefferson University
Locations (2):
- United States (2):
  - Kennedy Health Systems- Cancer Center, Sewell, New Jersey
  - Thomas Jefferson University Hopsital, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No